CLINICAL TRIAL: NCT02469701
Title: Nivolumab and Ablation For Patients With Advanced Non-Small Cell Lung Cancer Progressing After at Least One Prior Therapy For Metastatic Disease: A Brown University Oncology Research Group Phase II Study
Brief Title: Advanced Non-Small Cell Lung Cancer Progressing After at Least One Prior Therapy For Metastatic Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: howard safran (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor-Investigator, howard safran, Prinicipal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 317
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; Metastatic Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab with ablation (Experimental): 3mg/kg IV over 60 minutes on Day 1 +/- 3 days every 2 weeks until progression for a maximum of 2 years.
  Either cryoablation or thermal ablation may be performed as per standard institutional policies.
  As of amendment # 7 submitted to sites November 17, 2017, the dosing for Nivolumab per the FDA guidance was amended to a flat dose of 240mg IV Q2 weeks. As of amendment #8 sent to sites February 22, 2017 the dose of Nivolumab was updated to 3 mg/kg with a maximum dose of 240 mg for patients with weights that would correlate to exceed that dose instead of a flat dose secondary to the standard institutional practice and the FDA guidance .
  Interventions: Drug: nivolumab and ablation

INTERVENTIONS:
Drug: nivolumab and ablation
  Other Names: Opdivo

SUMMARY:
Nivolumab releases the inhibition of the immune system against human cancers. Dramatic and sustained activity has been observed in advanced lung cancer. Ablation may stimulate the immune system by exposing new tumor antigens. Since tumors that express PD-L1 may be more likely to respond to nivolumab, if ablation increases PD-L1 expression (which has not been studied) this treatment may enhance the activity of nivolumab at both the treated site and in other, non-treated, tumors. Ablation is already an FDA approved treatment for cancer. Nivolumab was recently FDA approved for second line treatment of advanced squamous cell NSCLC. The goal of the study will be to determine if the combination of nivolumab and ablation has higher systemic activity than previously reported with nivolumab alone.

DETAILED DESCRIPTION:
See summary above

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed NSCLC
* Stage IIIB or stage IV.
* Patient to meet either criterion A or B:

A) Progression after at least 1 line of systemic treatment (IV or oral) for metastatic or locally advanced disease. Must provide documentation systemic treatment was for either locally advanced or metastatic and also scan or assessment to show progression. Radiation does not count as 1 line.

B) Patients progressing within 6 months of completion of neoadjuvant or adjuvant chemotherapy are also eligible without having treatment for metastatic disease (for example patient with stage I disease undergoes resection, receives systemic chemotherapy and then progresses to the liver (now stage IV) within 6 months of chemotherapy). Radiation does not count as 1 line.

* Ablation for advanced lung cancer is being considered by the treating physician for treatment or prevention of symptoms such as pain, bleeding or obstruction- Documentation is required in writing by MD for this criterion.
* At least 1 site of measurable disease that will not be treated with ablation. Sites to send confirmation on which lesion of measurable disease will not be ablated for tracking of response.
* At least 3 weeks since prior chemotherapy and radiation therapy
* No brain metastases except for patients whose metastases have been removed by surgical resection or have had stereotactic radiation or gamma knife with no evidence of active disease on MRI within 28 days of starting treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Life expectancy of at least 12 weeks.
* Required entry laboratory parameters within 14 days of study entry: Granulocytes ≥ 1000/µl; platelet count ≥75,000/µl; absolute lymphocyte count ≥ 500/ µl; Creatinine ≤ 1.5x upper limit normal mg/dl; Bilirubin < 1.5x upper limit normal; AST ≤ 3 x upper limit of normal.
* Age > 18 years
* Men and women of childbearing potential enrolled in this study must agree to use adequate barrier birth control measures during the course of the study and up to 2 months after.
* Written informed consent.

Exclusion Criteria:

* Patients with a history of clinically significant chronic autoimmune disease
* Prior therapy with antibodies that modulate T-cell function defined as anti-CTLA-4, anti-PD-1, and anti-PD-L1
* Conditions currently requiring immunosuppressive medications
* Known history of HIV or hepatitis B or C
* Bleeding diathesis or coagulopathy that in the investigators opinion would prevent ablation from being safely performed.
* Patients with unstable angina (anginal symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* History of organ allograft even if not taking immunosuppressive medications
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab With Ablation: 3mg/kg IV over 60 minutes on Day 1 +/- 3 days every 2 weeks until progression for a maximum of 2 years.
  Either cryoablation or thermal ablation may be performed as per standard institutional policies
  nivolumab and ablation
  As of amendment # 7 submitted to sites November 17, 2017, the dosing for Nivolumab per the FDA guidance was amended to a flat dose of 240mg IV Q2 weeks. As of amendment #8 sent to sites February 22, 2017 the dose of Nivolumab was updated to 3 mg/kg with a maximum dose of 240 mg for patients with weights that would correlate to exceed that dose instead of a flat dose secondary to the standard institutional practice and the FDA guidance .
Period: Overall Study
Arm/Group | Nivolumab With Ablation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab With Ablation: 3mg/kg IV over 60 minutes on Day 1 +/- 3 days every 2 weeks until progression for a maximum of 2 years.
  Either cryoablation or thermal ablation may be performed as per standard institutional policies
  nivolumab and ablation
Arm/Group | Nivolumab With Ablation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of the Combination of Ablation and the PD-1 Inhibitor Nivolumab for Patients With Non-small Cell Lung Cancer (NSCLC) Who Have Progressed Following at Least 1 Prior Chemotherapy Regimen for Metastatic or Locally Advanced Disease.
Description: Assessment of tumor response by scan 12 weeks post the first dose of Nivolumab and approximately every 12 weeks after. Post progression by RECIST a 1 month confirmatory scan will be done and that will be the indicator of Progression.
Time Frame: Up to 5 years.
Population: Number of patients that were not known to Progress
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab With Ablation
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were required to be captured and reported from when the patient signed consent to 4 weeks post last dose of drug or until the subject withdraws consent from study participation (declines participation) or at the time patient becomes a screen failure, whichever occurs first.
Description: SAE capture includes a total of 6 initial medwatches effecting 5 patients (some gradable events within the medwtach may have occurred with multiple patients as outlined below in the affected/at risk table). Additional reports submitted to the FDA include follow up information regarding discharge, change of admission terms and administrative changes made to the report previously submitted.
Arm/Group | Nivolumab With Ablation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab With Ablation (N=10)
Sepsis, Pneumonia, Respiratory Failure (Investigations) | 1 (1)
Sepsis (Investigations) | 1 (1)
Myocardial Infarction, Respiratory Failure (Investigations) | 1 (1)
Spinal Fracture (Investigations) | 1 (1)
Fracture Rib (Investigations) | 1 (1)
Atrial Fibrillation (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab With Ablation (N=10)
agitation (Investigations) | 1 (1)
AKI (Investigations) | 1 (1)
Albumin (Investigations) | 5 (5)
ALK PHOS (ALP) (Investigations) | 3 (3)
allergic rhinitis (Investigations) | 2 (2)
ALT (Investigations) | 2 (2)
Anorexia (Investigations) | 6 (6)
anxiety (Investigations) | 2 (2)
apnea (Investigations) | 1 (1)
arthralgia (r shoulder, knee) (Investigations) | 3 (3)
Ascites (Investigations) | 1 (1)
Aspiration (Investigations) | 1 (1)
AST (Investigations) | 3 (3)
Reproductive system other : BPH (Investigations) | 1 (1)
CA (Investigations) | 3 (3)
chills/sweats (Investigations) | 3 (3)
confusion (Investigations) | 2 (2)
Congestive heart failure (Investigations) | 1 (1)
Constipation (Investigations) | 3 (3)
cough (productive cough) (Investigations) | 4 (4)
CR (Investigations) | 3 (3)
Dehydration (Investigations) | 3 (3)
Delirium (Investigations) | 2 (2)
depression (Investigations) | 1 (1)
Diarrhea (Investigations) | 3 (3)
Dizziness (Investigations) | 3 (3)
Dry eyes (Investigations) | 1 (1)
Dry mouth (Investigations) | 1 (1)
Dry skin (Investigations) | 1 (1)
Dysphagia (Investigations) | 2 (2)
dyspnea (Investigations) | 4 (4)
edema (limbs, bilateral lower extremity) (Investigations) | 2 (2)
Eye disorder other (double vision) (Investigations) | 1 (1)
Fatigue (Investigations) | 6 (6)
fever (Investigations) | 2 (2)
Fracture (spinal, rib) (Investigations) | 1 (1)
gait disturbance (Investigations) | 1 (1)
Glucose (Investigations) | 1 (1)
Headache (Investigations) | 2 (2)
HGB/ANEMIA (Investigations) | 8 (8)
HTN (Investigations) | 5 (5)
Hypotension (Investigations) | 2 (2)
Hypothyroidism (Investigations) | 1 (1)
hypoxia (Investigations) | 3 (3)
Infection and Infestations other ( sinus) (Investigations) | 1 (1)
INR (Investigations) | 4 (4)
insomnia (Investigations) | 2 (2)
K (Investigations) | 1 (1)
Lethargy (Investigations) | 1 (1)
Lymph (Investigations) | 5 (5)
Malaise (Investigations) | 1 (1)
MG (Investigations) | 1 (1)
muscle weakness (Investigations) | 2 (2)
Musculoskeletal other (soreness, trap spasm, impaired balance ) (Investigations) | 3 (3)
(Investigations) | 10 (10)
Nausea (Investigations) | 2 (2)
Neuropathy (Investigations) | 1 (1)
Pain -non cardiac various locations (Investigations) | 10 (10)
Palpitations (Investigations) | 1 (1)
Paresthesia (Investigations) | 1 (1)
pericardial effusion (Investigations) | 1 (1)
Pleural effusion (Investigations) | 5 (5)
PLT (Investigations) | 2 (2)
pneumonia (infection other) (Investigations) | 1 (1)
PO4 /PHOS (Investigations) | 3 (3)
Pruritus (Investigations) | 2 (2)
Pulmonary edema (Investigations) | 1 (1)
Rash (Investigations) | 2 (2)
Renal and Urinary disorders other(difficulty urinating ) (Investigations) | 1 (1)
Respiratory other (Hemoptysis) (Investigations) | 2 (2)
Restlessness (Investigations) | 1 (1)
Sore throat (Investigations) | 1 (1)
tachycardia (Investigations) | 1 (1)
Thromboembolic event (Investigations) | 1 (1)
Tinnitus (ear) (Investigations) | 1 (1)
Tremor (Investigations) | 1 (1)
Troponin I (Investigations) | 1 (1)
urinary frequency (Investigations) | 1 (1)
Vomit (Investigations) | 3 (3)
weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (5)
Wheezing (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02469701/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02469701/SAP_002.pdf